CLINICAL TRIAL: NCT01717963
Title: Optimal Prevention of Overdose Deaths and Opioid Relapse Following Discharge: A Multi-Center RCT of Naltrexone Versus Buprenorphine in Norway
Brief Title: Naltrexone vs Buprenorphine-Naloxone for Opioid Dependence in Norway
Acronym: NTX-SBX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); The Royal Norwegian Ministry of Health (Other); Norwegian Institute of Public Health (Other Government); Oslo University Hospital (Other); University Hospital, Akershus (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); The Hospital of Vestfold (Other); Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Lars Tanum, National Coordinating Investigator (PI), University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-002858-31; 204725-1 (Other Grant/Funding Number: Norwegian Research Council)
Record Dates: First submitted 2012-10-28; First posted 2012-10-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone intramuscular suspension (Experimental): Extended release naltrexone injections 380mg
  Interventions: Drug: Naltrexone intramuscular suspension
- Buprenorphine-naloxone (Active Comparator): Flexible oral dose 4-24 mg daily
  Interventions: Drug: Buprenorphine-naloxone

INTERVENTIONS:
Drug: Naltrexone intramuscular suspension — A standard dosage of 380 mg / month of naltrexone intramuscular suspension will be administered
  Other Names: Long-acting naltrexone; Extended-release naltrexone; XR-NTX; Vivitrol
  Arms: Naltrexone intramuscular suspension
Drug: Buprenorphine-naloxone — Buprenorphine-naloxone is administered daily and provided in accordance with existing guidelines for OMT in Norway (treatment-as-usual).
  Other Names: Suboxone
  Arms: Buprenorphine-naloxone

SUMMARY:
Persons dependent on opioids like heroin, morphine, or codeine have a high risk of relapse, overdose and overdose death. This risk is elevated even further following discharge from treatment or correctional institutions where patients have been detoxified. At the moment, state-of-the-art treatment is based on maintaining the dependence on opioids by daily intake of opioid medications like methadone or buprenorphine. Recently, a medication containing the blocking agent naltrexone was approved in the US; this does not maintain dependence but instead blocks heroin and other opioids for 28 days after intramuscular administration. This study will conduct a 12-week randomized comparison of naltrexone intramuscular suspension (XL-NTX) with daily buprenorphine-naloxone in OMT. Medication will start preceding discharge from a treatment or correctional facility to participating catchment regions in Norway. The main hypotheses are that XL-NTX will do equally well as - or better than - OMT on the proportion of biological samples negative for opioids, retention, self-reported use of alcohol and illicit drugs. Following the 12-week randomized period, there will be a 36-week period where participants can receive the study medication of their choice. After the end of the study, data from national registry databases can be collected for a further 12 months on outcomes such as recidivism, mortality and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependence (DSM-IV TR)
* Age 18 or above
* Applied & Approved for Norway's national OMT program
* Discharge within 30 days of inclusion from a controlled environment; e.g. inpatient treatment or correctional (prison) facility
* Voluntarily seeking treatment for opioid dependence

Exclusion Criteria:

* Pregnant or breast-feeding
* Acute or recurring severe psychiatric disorder, e.g. psychosis, suicidality
* Serious debilitation of liver or renal function (e.g. Child-Pugh level C)
* Use of excluded medication
* Known intolerance to study drugs or their ingredients
* Employment in firm manufacturing one of the study drugs or close relation to such person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08-31 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Number of biological samples negative/positive for opioid agonists | Week 1-12 post discharge
Retention | Week 1-12 post discharge
Days of use or abstinence from opioids | Week 1-12 post discharge

SECONDARY OUTCOMES:
Use of other substances of abuse | Week 1-48
Mental health | Week 1-12 or 1-48
  Self-reported mental health
Somatic health | Week 1-12 or 1-48 post discharge
  Self-reported and/or assessed by study personnel
Psychosocial problems | Week 1-12, Week 1-48, & Wk 49-100
  Psychosocial problems like recidivism, employment, family problems. Self-reported or registry-based.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Tanum, MD, PhD, Principal Investigator — University of Oslo
Locations (5):
- Norway (5):
  - Akershus University Hospital, Oslo, Akershus
  - Haukeland University Hospital, Bergen, Hordaland
  - Stavanger University Hospital, Stavanger, Rogaland
  - Vestfold Hospital Trust, Tønsberg, Vestfold
  - Oslo University Hospital, Avdeling for Rus og Avhengighet, Oslo

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Solli KK, Benth JS, Digranes LCW, Holtan L, Kunoe N, Tanum L. Changes in mental health during long-term treatment with extended-release naltrexone: A 3-year clinical study of opioid dependent individuals. Contemp Clin Trials. 2025 May;152:107861. doi: 10.1016/j.cct.2025.107861. Epub 2025 Feb 21. PMID 39987958
- [Derived] Opheim A, Benth JS, Solli KK, Kloster PS, Fadnes LT, Kunoe N, Gaulen Z, Tanum L. Risk of relapse to non-opioid addictive substances among opioid dependent patients treated with an opioid receptor antagonist or a partial agonist: A randomized clinical trial. Contemp Clin Trials. 2023 Dec;135:107360. doi: 10.1016/j.cct.2023.107360. Epub 2023 Oct 19. PMID 37865138
- [Derived] Opheim A, Gaulen Z, Solli KK, Latif ZE, Fadnes LT, Benth JS, Kunoe N, Tanum L. Risk of Relapse Among Opioid-Dependent Patients Treated With Extended-Release Naltrexone or Buprenorphine-Naloxone: A Randomized Clinical Trial. Am J Addict. 2021 Sep;30(5):453-460. doi: 10.1111/ajad.13151. PMID 34487395
- [Derived] Latif ZE, Solli KK, Opheim A, Kunoe N, Benth JS, Krajci P, Sharma-Haase K, Tanum L. No increased pain among opioid-dependent individuals treated with extended-release naltrexone or buprenorphine-naloxone: A 3-month randomized study and 9-month open-treatment follow-up study. Am J Addict. 2019 Feb;28(2):77-85. doi: 10.1111/ajad.12859. Epub 2019 Jan 31. PMID 30701613
- [Derived] Latif ZE, Saltyte Benth J, Solli KK, Opheim A, Kunoe N, Krajci P, Sharma-Haase K, Tanum L. Anxiety, Depression, and Insomnia Among Adults With Opioid Dependence Treated With Extended-Release Naltrexone vs Buprenorphine-Naloxone: A Randomized Clinical Trial and Follow-up Study. JAMA Psychiatry. 2019 Feb 1;76(2):127-134. doi: 10.1001/jamapsychiatry.2018.3537. PMID 30566177
- [Derived] Solli KK, Latif ZE, Opheim A, Krajci P, Sharma-Haase K, Benth JS, Tanum L, Kunoe N. Effectiveness, safety and feasibility of extended-release naltrexone for opioid dependence: a 9-month follow-up to a 3-month randomized trial. Addiction. 2018 Oct;113(10):1840-1849. doi: 10.1111/add.14278. Epub 2018 Jun 22. PMID 29806872
- [Derived] Tanum L, Solli KK, Latif ZE, Benth JS, Opheim A, Sharma-Haase K, Krajci P, Kunoe N. Effectiveness of Injectable Extended-Release Naltrexone vs Daily Buprenorphine-Naloxone for Opioid Dependence: A Randomized Clinical Noninferiority Trial. JAMA Psychiatry. 2017 Dec 1;74(12):1197-1205. doi: 10.1001/jamapsychiatry.2017.3206. PMID 29049469
- [Derived] Kunoe N, Opheim A, Solli KK, Gaulen Z, Sharma-Haase K, Latif ZE, Tanum L. Design of a randomized controlled trial of extended-release naltrexone versus daily buprenorphine-naloxone for opioid dependence in Norway (NTX-SBX). BMC Pharmacol Toxicol. 2016 Apr 28;17(1):18. doi: 10.1186/s40360-016-0061-1. PMID 27121539
- See also: Webpage of the study Sponsor: The Norwegian Centre for Addiction Research, Univ of Oslo — http://www.seraf.uio.no/